CLINICAL TRIAL: NCT03766750
Title: Randomized, Double-blind, Multicenter, National, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Lima Association in the Control of Type II Diabetes Mellitus
Brief Title: Efficacy and Safety of Lima Association in the Control of Type II Diabetes Mellitus.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS0318-LIMA
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — Linagliptin; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LIMA (Experimental)
  Interventions: Drug: LIMA association
- Tradjenta® (Active Comparator)
  Interventions: Drug: Tradjenta
- Forxiga® (Active Comparator)
  Interventions: Drug: Forxiga

INTERVENTIONS:
Drug: LIMA association — 1 coated tablet, oral, once a day.
  Other Names: EMS association
  Arms: LIMA
Drug: Tradjenta — 1 coated tablet, oral, once a day.
  Other Names: Linagliptin 5 mg
  Arms: Tradjenta®
Drug: Forxiga — 1 coated tablet, oral, once a day.
  Other Names: Dapagliflozin 10 mg
  Arms: Forxiga®

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Lima association in the control of type 2 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Participants of both sexes, aged 18 years or more;
* Participants presenting the diagnosis of type II diabetes mellitus, which have already received previous dietary and physical exercise guidance, who are not receiving any antidiabetic treatment, defined as never taking any antidiabetic medication, or in antidiabetic therapy after being subjected to a washout period;
* Treatment-naive participants with HbA1c between 7.5% and 10.5% and pretreated patients with HbA1c between 7,5% and 9,5% at the screening visit;
* Patients with HbA1c between 7.5% and 10.5% at the randomization visit;
* Participants with BMI (body mass index) > 19 Kg/m2 and ≤ 45 Kg/m2.
* Signed consent.

Exclusion Criteria:

* Any clinical and laboratory findings that, in the judgment of the investigator, may interfere with the safety of research participants;
* History of alcohol abuse or illicit drug use;
* Participation in clinical trial in the year prior to this study.
* Fasting glycemia above 300 mg/dL;
* Risk factors for severe volume depletion;
* Diuretic use less than 60 days, except for spironolactone;
* History of diabetic ketoacidosis;
* Medical history of acute coronary syndrome, stroke or transient ischemic attack within 3 months prior to informed consent;
* Impaired hepatic function;
* Impaired renal function and end stage renal disease;
* Bariatric surgery in the last two years and/ or other gastrointestinal surgeries;
* Current medical history of cancer and/ or cancer treatment in the last 5 years;
* Medical history of blood dyscrasia or any other hemolytic disorders;
* Medical history of pancreatitis and chronic pancreatitis;
* Treatment with anti-obesity drugs for less than 2 months or with dose change in the last 2 months;
* Current and prolonged treatment for more than 15 days with systemic steroids at the moment of informed consent;
* Any other uncontrolled endocrine disorder, except type 2 diabetes mellitus;
* History hypersensitivity to the active ingredients used in the study;
* Pregnancy or risk of pregnancy and lactating patients;
* Systemic disease that is not controlled and can put the participant at risk;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Reduction of glycated hemoglobin levels measured between the first visit and the last visit. | 120 days

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded during the study. | 210 days